CLINICAL TRIAL: NCT04562116
Title: An Open-label Drug-Drug Interaction Study to Assess the Effects of Nemolizumab on Cytochrome P450 Substrates in Subjects With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study to Assess the Effects of Nemolizumab on Cytochrome P450 Substrates in Participants With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RD.06.SPR.201593
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — nemolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CYP 450 Substrates plus Nemolizumab (Experimental): Participants will receive 1 single oral dose of selected, commercially available, cytochrome P450 substrates (CYP450-S) on Day 1 and after a 1-week washout period, participants will receive a 60 milligram (mg) loading dose of nemolizumab via 2 consecutive subcutaneous (SC) 30-mg injections at the Week 1 visit, followed by a single 30-mg injection once in every 4 weeks (Q4W) at Week 5 and Week 9. Participants will receive a second oral dosing of CYP450-S at Week 10.
  Interventions: Drug: Nemolizumab; Drug: CYP 450 Substrates

INTERVENTIONS:
Drug: Nemolizumab — Nemolizumab 30 mg will be administered as SC injections.
  Other Names: CD14152
Drug: CYP 450 Substrates — CYP substrates (Caffeine, Warfarin Sodium, Midazolam, Omeprazole, and Metoprolol Tartrate) will administered orally at Week 0 (Day 1) and Week 10 as per the commercially available prescribing information.

SUMMARY:
The purpose of this study is to evaluate the effect of nemolizumab (CD14152) on the pharmacokinetics (PK) of a drug "cocktail" representative of CYP450 (CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A4/5 sensitive index substrates) in adult participants with moderate to- severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Chronic atopic dermatitis (AD) for at least 2 years before the screening visit, and confirmed according to American Academy of Dermatology Consensus Criteria at the time of the screening visit
* Eczema Area and Severity Index (EASI) score greater than or equal to (>=) 16 at both the screening and baseline visits
* IGA score >= 3 (based on the Investigator's Global Assessment [IGA] scale ranging from 0 to 4, in which 3 is moderate and 4 is severe) at both the screening and baseline visits
* AD involvement >=10 percent (%) of body surface area (BSA) at both the screening and baseline visits
* Peak (maximum) pruritus numeric rating scale (PP NRS) score of at least 4.0 at both the screening and baseline visit
* Documented recent history (within 6 months before the screening visit) of inadequate response to topical medications (topical corticosteroid [TCS] with or without topical calcineurin inhibitor [TCI])

Exclusion Criteria:

* Body weight less than (<) 45 kilogram (kg)
* Participants meeting 1 or more of the following criteria at screening or baseline: (a) Had an exacerbation of asthma requiring hospitalization in the preceding 12 months; (b) Reporting asthma that has not been well-controlled in the previous 3 months; (c) Asthma Control Test (ACT) <= 19 (for those with a history of asthma); (d) Peak expiratory flow < 80% of the predicted value
* Participants with a current medical history of chronic obstructive pulmonary disease and/or chronic bronchitis
* Cutaneous infection within 1 week prior to the baseline visit, any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics or antifungals within 2 weeks prior to the baseline visit, or any confirmed or suspected coronavirus disease (COVID)-19 infection within 2 weeks before the screening or baseline visit. Participants may be rescreened once the infection has resolved. Resolution of COVID-19 infection can be confirmed by recovery assessment methods
* Requiring rescue therapy for AD during the screening period or expected to require systemic rescue therapy during the treatment period
* Positive serology results (hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb], hepatitis C antibody, or human immunodeficiency virus antibody) at the screening visit
* Treatment with systemic immunosuppressive/immunomodulating drugs and/or systemic corticosteroid within 4 weeks prior to Screening
* Known active or latent tuberculosis
* Treatment with Biologics and their biosimilars within 8 weeks from Screening
* Use of Phototherapy or tanning beds within 4 weeks from Screening
* Use of medication known as inducer, inhibitor, or competitive substrate of one or more of the following cytochrome (CYP) enzymes: CYP3A4/5, CYP2C19, CYP2C9, CYD2D6, and CYP1A2 within 2 weeks from Screening
* Treatment with Midazolam, Omeprazole, Warfarin Sodium, Metoprolol Tartrate within 2 weeks from Screening
* History of hypersensitivity or intolerance to CYP substrates and their excipients
* Participants for whom administration of the CYP substrates provided in this study is contraindicated or medically inadvisable
* Participants with international normalized ratio (INR) > 1.5
* Consumption of any 1 or more of the following food items and/or beverages within 1 week prior to baseline: Grapefruit or grapefruit juice, apple or apple juice, orange or orange juice, lemons or lemon juice, limes or lime juice, cranberries or cranberry juice; Vegetables from the mustard green family (eg, broccoli, kale); Charbroiled meats; Beverages, foods, or drugs containing caffeine
* History of or current confounding skin condition
* Current smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - 8894 Galderma Investigational Site, North Hollywood, California
  - 9954 Galderma Investigational Site, Hallandale, Florida
  - 9923 Galderma Investigational Site, Miami, Florida
  - 8030 Galderma Investigational Site, Raleigh, North Carolina
  - 8076 Galderma Investigational Site, Austin, Texas
- 5952 Galderma Investigational Site, Sofia, Bulgaria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 sites in the United States and Bulgaria from 08 December 2021 to 07 June 2023.
Pre-assignment Details: A total of 48 participants were screened, out of which 17 participants were enrolled in this study and 16 participants received at least 1 dose of nemolizumab.
Groups:
- CYP 450 Substrates Plus Nemolizumab: Participants received a single oral dose of selected, commercially available, cytochrome P450 substrates (CYP450-S) (caffeine 100 milligrams [mg], warfarin sodium 10 mg, midazolam 2 mg, omeprazole 20 mg, and metoprolol tartrate 100 mg) on Day 1. After a 1-week washout period, participants received a 60 mg loading dose of nemolizumab via 2 consecutive subcutaneous (SC) 30-mg injections at the Week 1 visit, followed by a single 30-mg injection once every 4 weeks (Q4W) at Week 5 and Week 9. Participants received a second oral dosing of CYP450-S at Week 10.
Period: Overall Study
Arm/Group | CYP 450 Substrates Plus Nemolizumab
Started | 17
Safety Population (Safety population included all participants who received at least 1 dose of Nemolizumab.) | 16
Completed | 13
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Enrolled population included all participants who signed the informed consent form and are enrolled in the study.
Groups:
- CYP 450 Substrates Plus Nemolizumab: Participants received a single oral dose of selected, commercially available, CYP450-S (caffeine 100 mg, warfarin sodium 10 mg, midazolam 2 mg, omeprazole 20 mg, and metoprolol tartrate 100 mg) on Day 1. After a 1-week washout period, participants received a 60 mg loading dose of nemolizumab via 2 consecutive SC 30-mg injections at the Week 1 visit, followed by a single 30-mg injection Q4W at Week 5 and Week 9. Participants received a second oral dosing of CYP450-S at Week 10.
Arm/Group | CYP 450 Substrates Plus Nemolizumab
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Area Under the Concentration-time Curve From Time Zero to Infinity (AUC[0-infinity]) of Each of the 5 Probe Drugs Before and After 9-week Nemolizumab Treatment
Description: AUC (0-infinity) was defined as AUC from time 0 to infinity, calculated as the sum of AUC (0-last) and C(last)/lambda(z); where C(last) was the last observed measurable (non-BQL) concentration; and lambda(z) was apparent terminal elimination rate constant. Probe drugs included Caffeine, Metoprolol Tartrate, Midazolam, Omeprazole and Warfarin Sodium. Change in AUC(0-infinity) of each of the 5 probe drugs before (Baseline) and after 9-week nemolizumab treatment is reported.
Time Frame: Baseline (before nemolizumab injection, at Week 0) and Week 10 (after nemolizumab injection): Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 72 and 120 hours post-dose
Population: Analysis was performed on the per-protocol population, which included all participants who completed the treatment period without any major protocol deviations or any other event that could render the probe drugs plasma concentration-time profiles unreliable. Here, number analyzed signifies the number of participants evaluable for each specified category.
Measure: Mean (Standard Deviation); unit: hour*microgram per liter
Groups:
- Before Nemolizumab Injections: Plasma pharmacokinetic parameters assessed before Nemolizumab injections i.e., at Baseline (Week 0).
- After Nemolizumab Injections: Plasma pharmacokinetic parameters assessed after 9 weeks of Nemolizumab injections i.e., at Week 10.
Arm/Group | Before Nemolizumab Injections | After Nemolizumab Injections
Number analyzed (Participants) | 14 | 14
hour*microgram per liter
  Caffeine | 27064 (16807) | 25281 (15146)
  Metoprolol Tartrate | 822 (698) | 845 (792)
  Midazolam | 27.7 (1.60) | 29.6 (15.0)
  Omeprazole: number analyzed (Participants) | 13 | 11
  Omeprazole | 932 (851) | 976 (715)
  Warfarin Sodium | 20268 (5261) | 20399 (4153)
Statistical Analysis 1: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Caffeine; Test type: Other; p = 0.5789, Mixed Models Analysis — A linear mixed-effect model was used to compare the natural log-transformed of the value, with substrate with or without Nemolizumab as the fixed effect and subject as a random effect; Ratio = 94.59, 90% CI 2-sided [79.57 to 112.45]
Statistical Analysis 2: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Metoprolol Tartrate; Test type: Other; p = 0.9468, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 99.34, 90% CI 2-sided [83.66 to 117.96]
Statistical Analysis 3: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Midazolam; Test type: Other; p = 0.1364, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 107.81, 90% CI 2-sided [99.14 to 117.24]
Statistical Analysis 4: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Omeprazole; Test type: Other; p = 0.1915, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 92.13, 90% CI 2-sided [82.85 to 102.44]
Statistical Analysis 5: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Warfarin Sodium; Test type: Other; p = 0.5059, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 101.67, 90% CI 2-sided [97.41 to 106.12]

2. Primary Outcome: Change in Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration (AUC [0-last]) of Each of the 5 Probe Drugs Before and After 9-week Nemolizumab Treatment
Description: AUC (0-last) was defined as AUC from time 0 to the time of the last measurable (non-BQL) concentration, calculated by linear-linear trapezoidal summation. Probe drugs included Caffeine, Metoprolol Tartrate, Midazolam, Omeprazole and Warfarin Sodium. Change of AUC(0-last) of each of the 5 probe drugs before (Baseline) and after 9-week nemolizumab treatment is reported.
Time Frame: as for outcome 1
Population: Analysis was performed on the per-protocol population, which included all participants who completed the treatment period without any major protocol deviations or any other event that could render the probe drugs plasma concentration-time profiles unreliable.
Measure: Mean (Standard Deviation); unit: hour*microgram per liter
Arm/Group | Before Nemolizumab Injections | After Nemolizumab Injections
Number analyzed (Participants) | 14 | 14
hour*microgram per liter
  Caffeine | 25294 (15633) | 23805 (13334)
  Metoprolol Tartrate | 803 (666) | 820 (742)
  Midazolam | 26.5 (12.4) | 28.5 (13.9)
  Omeprazole | 892 (825) | 796 (718)
  Warfarin Sodium | 18034 (4100) | 18068 (3470)
Statistical Analysis 1: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Caffeine; Test type: Other; p = 0.6665, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 95.82, 90% CI 2-sided [80.72 to 113.75]
Statistical Analysis 2: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Metoprolol Tartrate; Test type: Other; p = 0.9316, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 99.15, 90% CI 2-sided [83.43 to 117.83]
Statistical Analysis 3: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Midazolam; Test type: Other; p = 0.1371, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 107.75, 90% CI 2-sided [99.12 to 117.13]
Statistical Analysis 4: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Omeprazole; Test type: Other; p = 0.0962, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 88.66, 90% CI 2-sided [78.72 to 99.85]
Statistical Analysis 5: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Warfarin Sodium; Test type: Other; p = 0.6807, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 100.81, 90% CI 2-sided [97.45 to 104.29]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Each of the 5 Probe Drugs Before and After 9-week Nemolizumab Treatment
Description: Cmax was defined as the maximum observed plasma concentration. Probe drugs included Caffeine, Metoprolol Tartrate, Midazolam, Omeprazole and Warfarin Sodium. Cmax of each of the 5 probe drugs before (Baseline) and after 9-week nemolizumab treatment is reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | Before Nemolizumab Injections | After Nemolizumab Injections
Number analyzed (Participants) | 14 | 14
micrograms per liter
  Caffeine | 3922 (1563) | 3688 (1512)
  Metoprolol Tartrate | 200 (131) | 187 (114)
  Midazolam | 12.8 (5.31) | 11.8 (4.09)
  Omeprazole | 374 (205) | 349 (290)
  Warfarin Sodium | 695 (159) | 651 (174)
Statistical Analysis 1: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Caffeine; Test type: Other; p = 0.3431, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 91.22, 90% CI 2-sided [77.30 to 107.63]
Statistical Analysis 2: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Metoprolol Tartrate; Test type: Other; p = 0.4277, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 91.05, 90% CI 2-sided [74.33 to 111.53]
Statistical Analysis 3: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Midazolam; Test type: Other; p = 0.4963, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 94.79, 90% CI 2-sided [82.80 to 108.52]
Statistical Analysis 4: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Omeprazole; Test type: Other; p = 0.1931, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 88.24, 90% CI 2-sided [75.08 to 103.70]
Statistical Analysis 5: Comparison: Before Nemolizumab Injections vs After Nemolizumab Injections; Warfarin Sodium; Test type: Other; p = 0.2960, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio = 92.94, 90% CI 2-sided [82.51 to 104.69]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), AEs of Special Interest (AESIs), and Serious AEs (SAEs)
Description: An AE is defined as any untoward medical occurrence in a study participant administered a medicinal product which does not necessarily have a causal relationship with this treatment. SAE is any untoward medical occurrence that at any dose may results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. A TEAE is defined as an AE that occurs on or after the first date of study drug(s) administration until the date of last study visit. An AESI is a noteworthy treatment-emergent event for the study drug that should be monitored closely and reported promptly.
Time Frame: Up to 24 weeks
Population: Analysis was performed on the safety population. The safety population included all participants who received at least 1 dose of nemolizumab.
Measure: Count of Participants; unit: Participants
Groups:
- CYP 450 Substrates Plus Nemolizumab: Participants received 1 single oral dose of selected, commercially available, CYP450-S on Day 1. After a 1-week washout period, participants received a 60 mg loading dose of nemolizumab via 2 consecutive SC 30-mg injections at the Week 1 visit, followed by a single 30-mg injection Q4W at Week 5 and Week 9. Participants received a second oral dosing of CYP450-S at Week 10.
Arm/Group | CYP 450 Substrates Plus Nemolizumab
Number analyzed (Participants) | 16
Participants
  TEAEs | 0
  AESIs | 0
  SAEs | 0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: Analysis was performed on safety population which included all participants who received at least 1 dose of nemolizumab.
Arm/Group | CYP 450 Substrates Plus Nemolizumab
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT04562116/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT04562116/SAP_001.pdf